CLINICAL TRIAL: NCT00433199
Title: A Multi-Center, Randomized, Double-Blind,Placebo-Controlled Efficacy and Safety Study of Testosterone Gel 1.62% for the Treatment of Hypogonadal Men
Brief Title: Testosterone Treatment for Hypogonadal Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Michael Miller, Pharm. D Project Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S176.3.104
Record Dates: First submitted 2007-02-08; First posted 2007-02-09 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2011-11

CONDITIONS: Hypogonadism
Keywords: Hypogonadism; Testosterone Deficiency
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- T-Gel 1.62% (Experimental): Testosterone (T) gel 1.62%
  Interventions: Drug: Testosterone (T) Gel 1.62%

INTERVENTIONS:
Drug: Testosterone (T) Gel 1.62% — Testosterone gel 1.62% contains 1.62% testosterone gel as active ingredient.
  Arms: T-Gel 1.62%
Drug: Placebo — Placebo Control
  Arms: Placebo

SUMMARY:
Demonstrate efficacy and safety of Testosterone Gel 1.62% for the treatment of hypogonadal men

ELIGIBILITY:
Inclusion Criteria:

* Low T males 18 - 80 years of age

Exclusion Criteria:

* Normal T levels
* Elevated Prostatic Specific Antigen (PSA)

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2007-02; Primary Completion 2007-10 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Abbott Products

REFERENCES:
- [Derived] Kaufman JM, Miller MG, Fitzpatrick S, McWhirter C, Brennan JJ. One-year efficacy and safety study of a 1.62% testosterone gel in hypogonadal men: results of a 182-day open-label extension of a 6-month double-blind study. J Sex Med. 2012 Apr;9(4):1149-61. doi: 10.1111/j.1743-6109.2011.02630.x. Epub 2012 Feb 9. PMID 22321357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in 63 centers in US from February 2007 to April 2007 in clinics. The study was designed with a double-blind period of 182 days on Placebo or Androgel 1.62% followed by an 182 days open-label period on Androgel 1.62%.
Pre-assignment Details: All subjects started at a daily dose of 2.50 g testosterone gel 1.62% or matching placebo on Day 1. Within 2 days of each of visits (D14, D28 and D42), the dose was titrated up or down in 1.25 g steps if necessary, based on pre-specified normal range criteria, by an unblinded reviewer. The minimum and maximum daily doses were 1.25 g and 5.0 g.
Groups:
- Placebo: Placebo comparator administered during the Double-Blind period only
- T-Gel 1.62%: Testosterone (T): daily dose of 2.50 g testosterone gel 1.62% administered during the Double-Blind period and the Open-Label period.
Period: Double-Blind Period
Arm/Group | Placebo | T-Gel 1.62%
Started | 40 | 234
Completed | 28 | 168
Not Completed | 12 | 66
Not completed — Adverse Event | 0 | 25
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 8 | 19
Not completed — Protocol Violation | 1 | 10
Not completed — Administrative | 1 | 5
Period: Open-Label Period
Arm/Group | Placebo | T-Gel 1.62%
Started | 0 | 219
Completed | 0 | 185
Not Completed | 0 | 34
Not completed — Adverse Event | 0 | 19
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 0 | 7
Not completed — Protocol Violation | 0 | 2
Not completed — Administrative | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | T-Gel 1.62% | Total
Number analyzed (Participants) | 37 | 214 | 251
Age, Customized [Number; unit: participants] — The Baseline analysis is presented on the Full analysis set.
  participants
    <45 years | 7 | 34 | 41
    45-54 years | 7 | 83 | 90
    55-64 years | 16 | 67 | 83
    >= 65 years | 7 | 30 | 37
Sex: Female, Male [Count of Participants; unit: Participants] — The Baseline analysis is presented on the Full analysis set.
  Participants
    Female | 0 | 0 | 0
    Male | 37 | 214 | 251
Region of Enrollment [Number; unit: participants] — The Baseline analysis is presented on the Full analysis set.
  participants
    United States | 37 | 214 | 251

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects on Testosterone Treatment Achieving Target Range for Testosterone Cav (Time-averaged Concentration Over the Dosing Interval of 24 Hours) on Day 112
Description: Cav results were required to fall within the normal range of 300-1000 ng/dL. Success in the study was defined as >=75% of subjects on active treatment within the normal serum testosterone concentration range of 300-1000 ng/dL. In addition, the lower bound of the 95% CI was to be not less than 65% based on the Day 112 Parmacokinetics (PK) results
Time Frame: Day 112
Population: The analysis was done on the Full analysis sample defined as the subjects who were included in the Safety Sample and who had data for at least one post-Baseline assessment of any efficacy measurement up to and including Day 182 (double-blind period). The number correspond to the number of subjects having a measurement at Day 112;
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- T-Gel 1.62%: Testosterone gel 1.62% given during the double-blind period.
- Placebo: Placebo Comparator given during the double-blind period.
Arm/Group | T-Gel 1.62% | Placebo
Number analyzed (Participants) | 179 | 27
Percentage of subjects | 81.6 [75.1 to 87.0] | 37.0 [19.4 to 57.6]

2. Secondary Outcome: Percentage of Subjects on Testosterone Treatment Achieving Target Range for Testosterone Cav (Time-averaged Concentration Over the Dosing Interval of 24 Hours) on Day 14
Description: Cav results were required to fall within the normal range of 300-1000 ng/dL at Day 14. Success was defined as >=75% of subjects on active treatment within the normal serum testosterone concentration range of 300-1000 ng/dL. In addition, the lower bound of the 95% CI was to be not less than 65% based on the Day 14 PK results
Time Frame: Day 14
Population: The analysis was done on the Full analysis set with patients included in the double-blind period with a measurement at Day 14.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | T-Gel 1.62% | Placebo
Number analyzed (Participants) | 210 | 37
Percentage of subjects | 65.7 [58.9 to 72.1] | 29.7 [15.9 to 47.0]

3. Secondary Outcome: Percentage of Subjects on Testosterone Treatment Achieving Target Range for Testosterone Cav (Time-averaged Concentration Over the Dosing Interval of 24 Hours) on Day 56
Description: Cav results were required to fall within the normal range of 300-1000 ng/dL at Day 56. Success was defined as >=75% of subjects on active treatment within the normal serum testosterone concentration range of 300-1000 ng/dL. In addition, the lower bound of the 95% CI was to be not less than 65% based on the Day 56 PK results
Time Frame: Day 56
Population: The analysis was done on the Full analysis set with patients included in the double-blind period with a measurement at Day 56.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | T-Gel 1.62% | Placebo
Number analyzed (Participants) | 183 | 32
Percentage of subjects | 82.5 [76.2 to 87.7] | 34.4 [18.6 to 53.2]

4. Secondary Outcome: Percentage of Subjects on Testosterone Treatment Achieving Target Range for Testosterone Cav (Time-averaged Concentration Over the Dosing Interval of 24 Hours) on Day 182
Description: Cav results were required to fall within the normal range of 300-1000 ng/dL at Day 182. Success was defined as >=75% of subjects on active treatment within the normal serum testosterone concentration range of 300-1000 ng/dL. In addition, the lower bound of the 95% CI was to be not less than 65% based on the Day 182 PK results.
Time Frame: Day 182
Population: The analysis was done on the Full analysis set with patients included in the double-blind period with a measurement at Day 182.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | T-Gel 1.62% | Placebo
Number analyzed (Participants) | 169 | 28
Percentage of subjects | 82.2 [75.6 to 87.7] | 28.6 [13.2 to 48.7]

5. Secondary Outcome: Percentage of Subjects Achieving Target Range for Testosterone Cav During the Open-label Period at Day 266.
Description: The success at Day 266 was defined as >=75% of subjects within the normal serum total testosterone concentration range of 300-1000 ng/dL. The Lower bounds of the 95% CI was to be not less than 65%.
Time Frame: Day 266
Population: The analysis was done on the Full analysis set with patients included in the open-label period with a measurement at Day 266.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Continuing Active T-Gel 1.62% (CA): Testosterone gel 1.62% given during the Double-Blind period and Testosterone gel 1.62% given during the Open-label period.
- Formerly Placebo (FP): Placebo group given during the Double-Blind period and Testosterone gel 1.62% given during the Open-label period.
- Combined (CA and FP): Testosterone gel 1.62% is given to all the subjects entering the Open-label period.
Arm/Group | Continuing Active T-Gel 1.62% (CA) | Formerly Placebo (FP) | Combined (CA and FP)
Number analyzed (Participants) | 139 | 26 | 165
Percentage of subjects | 78.4 [70.6 to 84.9] | 69.2 [48.2 to 85.7] | 77.0 [69.8 to 83.2]

6. Secondary Outcome: Percentage of Subjects Achieving Target Range for Testosterone Cav During the Open-label Period at Day 364.
Description: The success at Day 364 was defined as >=75% of subjects within the normal serum total testosterone concentration range of 300-1000 ng/dL. The Lower bounds of the 95% CI was to be not less than 65%.
Time Frame: Day 364
Population: The analysis was done on the Full analysis set with patients included in the open-label period with a measurement at Day 364.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Formerly Placebo (FP): Placebo given during the Double-blind period and Testosterone gel 1.62% given during the Open-label period.
Arm/Group | Continuing Active T-Gel 1.62% (CA) | Formerly Placebo (FP) | Combined (CA and FP)
Number analyzed (Participants) | 136 | 23 | 159
Percentage of subjects | 77.9 [70.0 to 84.6] | 87.0 [66.4 to 97.2] | 79.2 [72.1 to 85.3]

ADVERSE EVENTS:
Time Frame: The adverse events presented were collected from start of drug treatment to the end of the double-blind treatment period (from Day 0 to Day 182).
Arm/Group | Placebo | T-Gel 1.62%
Serious Adverse Events (participants affected / at risk) | 1/40 | 5/234
Other Adverse Events (participants affected / at risk) | 5/40 | 47/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | T-Gel 1.62% (N=234)
Myocardial infarction (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pituitary Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spinal cord and nerve root disorders (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | T-Gel 1.62% (N=234)
Bacterial infections NEC (Infections and infestations) | 2 | 0
Upper respiratory tract infections (Infections and infestations) | 2 | 20
Cell marker procedures (Investigations) | 0 | 26
Headaches NEC (Nervous system disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At 60 days prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the Site shall provide to Sponsor a copy and allow Sponsor 60 days to review and comment.